CLINICAL TRIAL: NCT05102149
Title: A Multi-center, Randomized, Double-Blinded, Parallel, Vildagliptin and Placebo-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of PB-201 in Treatment-naive Patients With Type 2 Diabetes Mellitus
Brief Title: Study to Evaluate the Safety and Efficacy of PB-201 in Treatment-naive Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB201303
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Lead-201; Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test arm (Experimental): PB-201: 100 mg each time, orally in the morning and evening respectively; Vildagliptin matched placebo: One tablet each time, orally in the morning and evening respectively;
  Interventions: Drug: PB-201; Drug: Vildagliptin matched placebo
- Vildagliptin arm (Active Comparator): Vildagliptin: 50 mg each time, orally in the morning and evening respectively; PB-201 matched placebo: One tablet each time, orally in the morning and evening respectively;
  Interventions: Drug: Vildagliptin; Drug: PB-201 matched placebo
- Placebo arm (Placebo Comparator): PB-201 matched placebo: One tablet each time, orally in the morning and evening respectively; Vildagliptin matched placebo: One tablet each time, orally in the morning and evening respectively;
  Interventions: Drug: PB-201 matched placebo; Drug: Vildagliptin matched placebo

INTERVENTIONS:
Drug: PB-201 — PB-201: 100 mg each time, orally in the morning and evening respectively;
  Arms: Test arm
Drug: Vildagliptin — Vildagliptin: 50 mg each time, orally in the morning and evening respectively;
  Arms: Vildagliptin arm
Drug: PB-201 matched placebo — PB-201 matched placebo: One tablet each time, orally in the morning and evening respectively;
  Arms: Placebo arm; Vildagliptin arm
Drug: Vildagliptin matched placebo — One tablet each time, orally in the morning and evening respectively;
  Arms: Placebo arm; Test arm

SUMMARY:
This is a multicenter, randomized, double-blind, parallel, Vildagliptin and Placebo-Controlled study to evaluate the efficacy and safety of oral administration of 100 mg of PB-201 in the morning and evening in treatmentnaive patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The study consists of a screening period of up to 2 weeks, a 4-week single-blind run-in period, a 24-week double-blinded treatment period, a 28-week extended treatment period, and a 2-week safety follow-up period.Eligible subjects will be enrolled in a 4-week single-blind run-in period with daily oral administration of 1 tablet of PB-201 matched placebo and 1 Vildagliptin matched placebo in the morning and evening respectively.After the end of the single-blind run-in period, subjects who meet the protocol enrollment requirements will be randomized in the proportion of 2:1:1 to receive double-blinded treatment for 24 weeks in three different treatment groups (test arm, Vildagliptin arm, or placebo arm).

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for this study:
* Males or females aged ≥18 years and ≤ 75 years at screening;
* Diagnosed T2DM patients who meet the diagnostic criteria for type 2 diabetes mellitus issued by WHO in 1999 (see Appendix 2 for diagnostic criteria of type 2 diabetes mellitus);
* Receive diet and exercise interventions for at least eight weeks before screening and do not receive any anti-diabetes medications within eight weeks before screening;
* The Glycosylated hemoglobin (HbA1c) must meet the following criteria:

  1. HbA1c ≥ 7.5% and ≤ 11.0% at screening (local laboratory);
  2. HbA1c ≥ 7.0% and ≤ 10.5% (central laboratory) prior to randomization (V3);
* Body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 40.0 kg/m2 at screening or prior to randomization (V3);
* Able to understand and willing to sign the written informed consent form (ICF) and follow the protocol.

Exclusion Criteria:

* Patients cannot be randomized if they meet any of the following criteria:
* Patients diagnosed with type 1 diabetes mellitus, diabetes due to pancreatic injury, or special type of diabetes due to other diseases (e.g., acromegaly or Cushing's syndrome);
* Patients who receive other glucokinase activators prior to screening or randomization;
* Patients who have acute diabetic complications such as diabetic ketoacidosis, lactic acidosis or hyperglycemia and hyperglycemic hyperosmolar status within six months before screening or prior to randomization;
* Patients who have severe chronic diabetic complications (such as proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot, etc.) within six months before screening.
* Patients who have two or more episodes of severe hypoglycemia within six months before screening, or who have had severe hypoglycemia prior to randomization since screening ;
* Patients who have hemorrhagic stroke or acute ischemic stroke within six months before screening or prior to randomization;
* Patients who have a history of acute or chronic pancreatitis at screening or prior to randomization;
* Patients who suffer from any serious gastrointestinal diseases (such as gastroparesis, inflammatory bowel disease, intestinal obstruction) that affect drug absorption within six months before screening or prior to randomization, or have underwent gastrointestinal operations that affect drug absorption (such as gastrectomy, gastroenterostomy or enterectomy, etc.);
* Patients who have severe trauma or serious infection that may affect glycaemic control within one month before screening or prior to randomization, such as bone fracture, pneumonia, etc.;
* Patients with any type of treated or untreated malignancy (whether cured or not) within five years before screening or prior to randomization. However, patients with cured basal cell carcinoma of the skin do not need to be excluded;
* Patients with thyroid dysfunction not controlled by stable drug dosage at screening or abnormalities of thyroid function test with clinically significant at screening and requiring medical treatment;
* Patients who have any of the following laboratory abnormalities at screening:

  1. Human immunodeficiency virus antibody or Treponema pallidum specific antibody positive;
  2. Hepatitis C antibody positive;
  3. Hepatitis B surface antigen is positive, and the result of hepatitis B virus DNA quantitative test is higher than the lower limit of the test reference range (Note: If the local laboratory cannot carry out quantitative detection of hepatitis B virus, the sample will be sent to the central laboratory.);
* Patients who have any disease at screening or prior to randomization that may cause hemolysis or red blood cell instability affecting HbA1c testing, such as hemolytic anemia;
* Subject who has participated in any drug or medical device clinical study within three months before screening or prior to randomization (except those who fail in screening or do not receive any trial drug);
* Patients who have a prior history of clearly diagnosed psychiatric disorders, unwilling or unable to fully understand and cooperate, or assessed by the investigator as unsuitable for participation in this clinical study;
* Patients who have a prior history of drinking [(>2 units of alcohol per day and >14 units of alcohol per week (one unit of alcohol corresponds to 150mL of grape wine or 350mL of beer or 50 mL of spirits)] or history of drug abuse;
* Patients who are known to be allergic or intolerant to the test drug or Vildagliptin or their excipients, or who have contraindications;
* Patients who have refractory urinary or genital infections within six months before screening, or are known to be allergic to Empagliflozin or its excipients;
* Female in pregnancy or lactation period;
* Partners of male subjects or female subjects who plan to become pregnant or who are unable or unwilling to use contraceptive methods required by the protocol from the signing of the informed consent form to 30 days after the last dose of the drug;
* The investigator judges that the subject is unable to comply with the protocol requirements, such as unable to adhere to diet and exercise treatment during the study, unable to take drugs and meals on time according to the protocol requirements, and unable to conduct self-monitoring of blood glucose (SMBG) in time and record;
* Other circumstances that, in the opinion of the investigator, are not appropriate for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 1,Week 25
  Change from baseline in HbA1c after 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD,PhD, Principal Investigator — Peking University People's Hospital
Locations (42):
- China (39):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Lu'an People's Hospital, Lu'an, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Handan First Hospital, Handan, Hebei
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Qiqihar, Qiqihar, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - The Third Hospital of Changsha, Changsha, Hunan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hunan
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Sir Run Run Hospital Nanjing Medical Universtiy, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Nantong First People's Hospital, Nantong, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Panjin LiaoHe Oil Field Gem Flower Hospital, Panjin, Liaoning
  - Tangdu Hospital, Air Force Medical University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Peace Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - The Third People's Hospital of Datong, Datong, Shanxi
  - Yan'an University Affiliated Hospital, Ya'an, Shanxi
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
- Hong Kong (2):
  - The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
  - The University of Hong Kong, Queen Mary Hospital, Hong Kong
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No